CLINICAL TRIAL: NCT02759172
Title: Suicide Risk Reduction in the Year Following Jail Release: the SPIRIT Trial (Suicide Prevention Intervention for At-Risk Individuals in Transition)
Brief Title: Suicide Prevention Intervention for At-Risk Individuals in Transition
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Jennifer E. Johnson, Principal Investigator, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01MH106660 (NIH)
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Suicide
Keywords: Suicide prevention; Jail
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safety Planning Intervention (Experimental): Brown and Stanley's Safety Planning Intervention (SPI) is a brief, adjunctive intervention designed to reduce subsequent suicidal behavior in high-risk populations. The core element of SPI is the collaborative development of the Safety Plan, which is a prioritized written list of coping strategies and supports that individuals can use during or preceding suicidal crises. In this study, safety planning will occur during pretrial jail detention, with telephone follow-up in the community to conduct risk assessment, review the Safety Plan, problem-solve obstacles to treatment, and assist with linkage to services.
  Interventions: Behavioral: Safety Planning Intervention
- Standard Care (No Intervention): Standard Care for pretrial jail detainees is assessment of risk and stabilization to the extent possible during their jail detention. No post-release community follow-up is typically provided. This study will augment standard care with regular assessment and emergency referral post-release, as well as provision of a list of community resources.

INTERVENTIONS:
Behavioral: Safety Planning Intervention — Brown and Stanley's Safety Planning Intervention (SPI) is a brief, adjunctive intervention designed to reduce subsequent suicidal behavior in high-risk populations. The core element of SPI is the collaborative development of the Safety Plan, which is a prioritized written list of coping strategies and supports that individuals can use during or preceding suicidal crises. In this study, safety planning will occur during pretrial jail detention, with telephone follow-up in the community to conduct risk assessment, review the Safety Plan, problem-solve obstacles to treatment, and assist with linkage to services.
  Other Names: SPI
  Arms: Safety Planning Intervention

SUMMARY:
The four year SPIRIT Trial, or Suicide Prevention Intervention for at-Risk Individuals in Transition, will recruit 800 pretrial jail detainees at risk for suicide. Each participant will be randomly assigned to today's standard care or to Safety Planning Intervention (SPI) method and then followed for one year after release. Outcomes include suicide events, suicide attempts and ideation, psychiatric symptoms, functioning, treatment utilization, problem-solving, belongingness, and cost-effectiveness.

DETAILED DESCRIPTION:
There were nearly 12 million admissions to US jails in 2012. Jailed individuals face a disproportionate risk for suicide. The time of arrest and jail detention represents an acute stressor that further exacerbates this risk. The epidemic of suicide during jail detention has been recognized. However, less attention has been paid to the high suicide risk and mortality in the months following jail release, as individuals re-enter their communities, are faced with financial, legal, and social stressors, and have increased access to lethal means (e.g., drugs, cars, firearms). Given that roughly 10% of all suicides in the U.S. with known circumstances occur following a recent criminal legal stressor (often arrest and jail detention), reducing suicide risk in the year after jail detention could have a noticeable impact on national suicide rates. Unlike prison, where individuals have already been sentenced and typically stay from months to years, most pretrial jail detainees are released within days. Therefore, brief interventions are required. Stanley and Brown's Safety Planning Intervention (SPI) is a brief, adjunctive suicide risk reduction intervention developed for suicidal patients presenting to urgent care settings. SPI incorporates evidence-based suicide risk reduction strategies in a low intensity, low cost intervention that can be delivered by a broad range of clinicians, making it scalable in the mental health resource-poor justice system. SPI reduces subsequent suicidal ideation and attempts among at-risk individuals in emergency rooms. However, there is no previous test of this intervention (or any other) for reducing suicidality following jail release. This RCT evaluates the effectiveness and cost-effectiveness of SPI for reducing suicide events (attempts, suicide behaviors, and suicide-related hospitalizations and emergency department visits) and attempts among 800 suicidal pretrial jail detainees from two jails in the year following jail release. It assesses critical mechanisms of suicide reduction in our target population: treatment utilization, suicide-related problem-solving, and belongingness. SPI will consist of safety planning during jail detention and follow-up phone sessions after jail release. Research with previously incarcerated individuals and with suicidal individuals in the community has shown that telephone follow-up intervention is feasible and powerful in building trust and reducing risk among these disenfranchised, isolated populations. This study will be the first randomized evaluation of a suicide prevention intervention in the vulnerable year after jail release. Beyond the human suffering and costs at an individual level, suicidal behavior incurs high economic costs in terms of health care costs and lost productivity. Jails are a catchment area for at-risk individuals at a time of high life stress and high suicide risk, providing an important opportunity for suicide prevention intervention, one that is currently being missed. This study will provide the data on costs and cost-adjusted outcomes that systems need to make informed decisions about adoption, speeding implementation. Thus, this study will contribute to knowledge about both mechanisms of action and system-level intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Unsentenced male and female pretrial jail detainees
* 18+ years of age
* at risk for suicide, operationalized as a response of "yes" on item 4 or greater on the initial 5 C-SSRS screening questions, indicating the presence of at least some active suicide ideation with some intent to act in the past month (i.e., individuals at higher risk, such as those who report intent with specific plan and/or suicide attempt/s in the last month, will also be included);
* speak and understand English well enough to understand questionnaires when they are read aloud.

Exclusion Criteria:

* expects to be sentenced and serve their sentence before being released to the community
* cannot provide the name and contact information of at least two locator persons
* does not have access to any telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, PhD, Principal Investigator — Michigan State University; Lauren Weinstock, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Genesee County Jail, Flint, Michigan
  - Rhode Island Department of Corrections, Cranston, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available through relevant NIH and NIJ repositories after the trial has ended.

REFERENCES:
- [Derived] Weinstock LM, Jones RN, Miller TR, Brown GK, Arias SA, Graves HR, Miller IW, Cerbo L, Rexroth J, Fitting H, Russell D, Kubiak S, Stein MD, Matkovic C, Yen S, Gaudiano BA, Johnson JE. Safety Planning vs Standard Care for Suicide Prevention After Pretrial Jail Detention: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543156. doi: 10.1001/jamanetworkopen.2025.43156. PMID 41212557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety Planning Intervention | Standard Care
Started | 402 | 398
Completed | 342 | 313
Not Completed | 60 | 85

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Planning Intervention | Standard Care | Total
Number analyzed (Participants) | 342 | 313 | 655
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.2) | 33.2 (10.5) | 33 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 84 | 182
  Male | 244 | 229 | 473
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 175 | 173 | 348
  Black or African American | 83 | 76 | 159
  American Indian or Alaskan Native | 39 | 32 | 71
  All other groups and not-specified | 45 | 32 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity | 49 | 38 | 87
  Non-Hispanic Ethnicity | 293 | 275 | 568

OUTCOME MEASURES:

1. Primary Outcome: Suicide Events
Description: Number of suicide events (a composite of attempts, behaviors, suicide-related hospitalizations, and suicide deaths) in the year following jail release. Events are identified through self-report, hospital records, and death records.
Time Frame: One year after jail release
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
number of events | 1.8 (3.4) | 3.0 (7.2)

2. Secondary Outcome: Suicide Attempts
Description: Number of suicide attempts using the Columbia (C-SSRS) criteria.
Time Frame: One year after release from jail
Measure: Mean (Standard Deviation); unit: Number of attempts
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
Number of attempts | 1 (2.7) | 2.1 (6.4)

3. Secondary Outcome: Weeks of Active Suicide Ideation
Description: Operationalized using the Longitudinal Interval Follow-Up Evaluation (LIFE)
Time Frame: One year after release from jail
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 312 | 282
weeks | 9 (11.5) | 10.9 (13.1)

4. Secondary Outcome: Severity of Suicide Ideation
Description: Columbia Suicide Severity Rating Scale (C-SSRS) Suicide Intensity Subscale score. Subscale scores range from 2 to 25, higher scores indicating more intense suicidal ideation.
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Deviation); unit: score on a subscale
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 312 | 283
score on a subscale | 15.2 (7.7) | 16.2 (7.1)

5. Secondary Outcome: Time to First Suicide Event
Time Frame: One year after release from jail
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
weeks | 7.4 (6.3) | 4.4 (3.8)

6. Secondary Outcome: Psychiatric Symptoms
Description: NIH's Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Cross-Cutting Measure total score. Scores range from 0 to 92, higher scores reflecting greater severity of psychiatric symptoms.
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 308 | 280
score on a scale | 44.1 (18.4) | 45 (19.3)

7. Secondary Outcome: Functioning
Description: Veterans RAND 12-Item Health Survey (VR-12) total score. Scores range from 0 to 100, higher scores indicating greater functioning.
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 308 | 280
score on a scale | 72 (18.9) | 72.3 (19.2)

8. Secondary Outcome: Treatment Utilization
Description: Number of outpatient mental health and substance use visits attended
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Error); unit: number of visits
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
number of visits | 9.02 (0.88) | 8.41 (0.86)

9. Secondary Outcome: Suicide-related Problem-solving
Description: Suicide-Related Coping Scale total score. Scores range from 0-68, higher scores indicating better suicide related coping.
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
score on a scale | 65.82 (0.66) | 65.39 (0.69)

10. Secondary Outcome: Belongingness
Description: Interpersonal Needs Questionnaire-12 (INQ-12) belongingness subscale score. Scores range from 0-54, higher scores indicating higher levels of thwarted belongingness.
Time Frame: Assessed 1, 4, 8, and 12 months after release from jail, 12 months reported.
Measure: Mean (Standard Error); unit: score on a subscale
Arm/Group | Safety Planning Intervention | Standard Care
Number analyzed (Participants) | 342 | 313
score on a subscale | 19.90 (0.77) | 20.08 (0.81)

ADVERSE EVENTS:
Time Frame: Assessed from consent through 1 year after release from jail, up to 27 months.
Arm/Group | Safety Planning Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 12/342 | 4/313
Serious Adverse Events (participants affected / at risk) | 177/342 | 159/313
Other Adverse Events (participants affected / at risk) | 70/342 | 69/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Planning Intervention (N=342) | Standard Care (N=313)
Suicide attempt (Psychiatric disorders) | 129 | 128 — Non-fatal suicide attempt
Inpatient hospitalization (Psychiatric disorders) | 82 | 72 — Suicide or potentially suicide related inpatient hospitalization
Death (Psychiatric disorders) | 12 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Planning Intervention (N=342) | Standard Care (N=313)
Non-suicidal self-injurious behavior (Psychiatric disorders) | 68 | 69
Distress during the assessment (General disorders) | 1 | 0
Access of confidential information by non-authorized person (Social circumstances) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02759172/Prot_SAP_000.pdf